The Effect of Synbiotic Tablet Usage on the Clinical and Biochemical

Parameters in Smokers and Nonsmokers with Gingivitis: A Randomized

**Placebo-Controlled Clinical Trial** 

**Document Date: February 27, 2018** 

## **Statistical Analysis**

The suitability of the normal distribution of the variables in our study was evaluated with graphical and Shapiro-Wilks test. The median (minimum, maximum) was used to display the descriptive statistics of variables identified as an abnormal distribution. Number (n) and percentage values were given to show the distribution of categorical variables like gender.

Kruskal-Wallis non-parametric analysis of variance was used to examine if there has been anydiscrepancy in the values of the clinical and biochemical measurements at baseline, 1st month and 2nd month. Bonferroni correction with the dual comparisons were made to determine the group causing variations in the variables found significant differences as result of Kruskal-Wallis test.

For comparing the clinical, biochemical and microbiological measurements at baseline, 1 month and 2 months in each group (T(+) T(-), C(+), C(-)) Friedman non-parametric repeated measures analysis of variance was used. Bonferroni correction double comparisons were made in variables determined statistically significant differences from the result of the Friedman test.

G\*Power pack program<sup>‡‡‡</sup> was used in order to determine the number of samples used in the study. For the width effect f: 0.25, type-I error probability  $\alpha$ :0.05, type-II error probability  $\beta$ : 0.05 and power: 0.95, at least 15 sampling units have been calculated to include in the study for each group. At least 5 subjects were added for each group considering the missing data that was deemed to occur during the course of follow-up. Sample size calculation was attempted based on the primary outcome measure.